CLINICAL TRIAL: NCT06712563
Title: Pooled Analysis of Multi-country, Open-label Single-arm, Non-interventional, Multi-center, Cohort Studies of Real-world Outcomes in New Users of Budesonide/Glycopyrronium/Formoterol (BGF) in Routine Care Setting
Brief Title: Pooled Analysis of Single-arm Studies of Budesonide/Glycopyrronium/Formoterol (BGF) in Routine Care Setting
Acronym: CHOROS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00084
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — budesonide-glycopyrrolate-formoterol fumarate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BGF Initiators: New initiators of BGF without prior BGF exposure
  Interventions: Drug: Budesonide/glycopyrrolate/formoterol fumarate

INTERVENTIONS:
Drug: Budesonide/glycopyrrolate/formoterol fumarate — Budesonide/glycopyrrolate/formoterol fumarate (BGF) is a triple fixed-dose combination therapy for adults with moderate to severe COPD who are not adequately treated by a combination of inhaled corticosteroids and long-acting beta-agonist (LABA), or LABA and long-acting muscarinic-antagonist
  Other Names: BGF, Breztri

SUMMARY:
The CHOROS pooled analysis is a retrospective secondary data use analysis of integrated individual participant data from a series of planned and on-going primary prospective, non-interventional, multi-center studies sponsored by AstraZeneca and conducted in the pulmonary/primary care practitioner setting in multiple countries and may include data from the following countries: United Kingdom, Germany, Italy, Greece, Japan, Canada and Romania.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe COPD and initiating BGF treatment according to the local prescribing guidance and as per their treating physician's recommendation
* Enrolled in on-going single-arm studies
* Provided consent for secondary use of data

Exclusion Criteria:

* Did not provide consent for secondary use of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD who are new initiators of BGF enrolled in several planned and on-going prospective, non-interventional single-arm studies. Eligible patients for the individual studies are those with moderate to severe COPD and initiating BGF treatment according to the local prescribing guidance and as per their treating physician's recommendation. Only patients that have signed an informed consent form (ICF) allowing the secondary use of their data will be eligible for the CHOROS pooled analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 12 weeks
  Compare self-reported COPD health status measured by COPD Assessment Test (CAT) at 12 weeks/3 months as compared to baseline in patients initiating treatment with BGF

SECONDARY OUTCOMES:
COPD Assessment Test | 4 weeks
  To compare self-reported COPD health status measured by CAT at 4 weeks/1 month as compared to baseline in patients initiating treatment with BGF
COPD Assessment Test | 52 weeks
  To compare self-reported COPD health status measured by CAT at 52 weeks/12 months as compared to baseline in patients initiating treatment with BGF
COPD Assessment Test Responder Rate | 12 weeks
  To describe the frequency and proportion of responders of the CAT questionnaire after 12 weeks/3 months of initiating treatment with BGF
Treatment Satisfaction Questionnaire for Medication (TSQM) | 12 weeks and 52 weeks
  To evaluate treatment satisfaction using Treatment Satisfaction Questionnaire for Medication (TSQM) after 12 weeks/3months and 52 weeks/12 months of initiating treatment with BGF
Annual rate of COPD exacerbations | 52 weeks
  To compare the annual rates of moderate and severe exacerbations for the follow-up period (up to 52 weeks/12 months) versus the baseline period (12 months prior to initiating BGF)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Pollack, MS, Principal Investigator — AstraZeneca
Locations (7):
- Research Site, Mississauga, Canada
- Research Site, Hamburg, Germany
- Research Site, Athens, Greece
- Research Site, Milan, Italy
- Research Site, Tokyo, Japan
- Research Site, Bucharest, Romania
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/